CLINICAL TRIAL: NCT05708066
Title: Aromatherapy With Lavender as Anxiolysis Prior to Cataracts Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never approved by the Albert Einstein College of Medicine IRB
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-13826
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Aromatherapy; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Aromatherapy Tab (Experimental): If part of the experimental group, participants will have the Bioesse lavender patch placed on the chest, according to manufacturer recommendations. After the lavender patch has been in place for 5 minutes, participants will receive the same visual analogue scale (VAS) anxiety questionnaire.
  Interventions: Other: Lavender Aromatherapy
- Non-scented Tab (Placebo Comparator): If part of the placebo comparator group, participants will have an unscented tab placed on the chest, according to manufacturer recommendations. Participants in this group will only receive the initial visual analogue scale (VAS) anxiety questionnaire.
  Interventions: Other: Non-scented Tab

INTERVENTIONS:
Other: Lavender Aromatherapy — Participants will have the Bioesse lavender patch placed on the chest, according to manufacturer recommendations.
  After the lavender patch has been in place for 5 minutes, the same VAS anxiety questionnaire will be provided
  Arms: Lavender Aromatherapy Tab
Other: Non-scented Tab — A non-scented tab will be placed on the participant's chest, according to manufacturer recommendations. Participants in this group will only receive the initial VAS anxiety questionnaire.
  Arms: Non-scented Tab

SUMMARY:
The purpose of this study is to assess the validity of lavender aromatherapy as a method of anxiolysis prior to a cataract surgery, and to see if this effect will extend intraoperatively to minimize patients' intraoperative medication requirements. The study team plans on enrolling 186 participants.

The investigator team hypothesizes that:

1. Participants will have a lower anxiety score after the intervention
2. Participants will require less intraoperative sedation medication compared to participants that did not have the lavender intervention.
3. A decrease in intraoperative medication requirements will lead to a faster discharge time

DETAILED DESCRIPTION:
All participants will arrive at the Hutchinson Campus on the morning of surgery. After nursing intake, participants will be consented into the study. Vital signs will be recorded, as is part of the typical nursing intake. After the consent is completed, participants will receive the visual analogue scale (VAS) anxiety questionnaire. Participants that are part of the experimental group will then have the Bioesse lavender patch placed on the chest, according to manufacturer recommendations. After the lavender has been in place for 5 minutes, the same VAS anxiety questionnaire will be provided for completion. The control subjects will only receive the initial VAS questionnaire.

After this, all participants will receive the same premedication, including fentanyl and midazolam prior to cataract surgery, and will have monitored anesthesia care (MAC) during the case.

In the second phase of the study, chart review will be completed to monitor the patients' intraoperative sedation requirements . Additionally, demographic data will be taken at this time, including age, race, and sex.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* ASA (American Society of Anesthesiology) score <=3
* Patients must be able to consent to participating in the study

Exclusion Criteria:

* ASA score >4
* Patients with a psychiatric diagnosis or who are on psychiatric medication
* Patients with a history of asthma
* Patients with an allergy to lavender
* Patients under an anesthetic plan that has been switched from local anesthesia with sedation to general anesthesia
* VAS score > 60 pre-operatively (high anxiety score)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Effect of lavender aromatherapy on anxiolysis | Based on intra-operative time
  Patient intra-operative data will be assessed to check dosage of midazolam and fentanyl between the placebo and intervention groups to see if lavender aromatherapy provides intra-operative anxiolysis cataracts surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Steinberg, DO, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center Hutchinson Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abend R, Dan O, Maoz K, Raz S, Bar-Haim Y. Reliability, validity and sensitivity of a computerized visual analog scale measuring state anxiety. J Behav Ther Exp Psychiatry. 2014 Dec;45(4):447-53. doi: 10.1016/j.jbtep.2014.06.004. Epub 2014 Jun 18. PMID 24978117
- [Background] Cho MY, Min ES, Hur MH, Lee MS. Effects of aromatherapy on the anxiety, vital signs, and sleep quality of percutaneous coronary intervention patients in intensive care units. Evid Based Complement Alternat Med. 2013;2013:381381. doi: 10.1155/2013/381381. Epub 2013 Feb 17. PMID 23476690
- [Background] Jaruzel CB, Gregoski M, Mueller M, Faircloth A, Kelechi T. Aromatherapy for Preoperative Anxiety: A Pilot Study. J Perianesth Nurs. 2019 Apr;34(2):259-264. doi: 10.1016/j.jopan.2018.05.007. Epub 2018 Sep 8. PMID 30205934
- [Background] Kang HJ, Nam ES, Lee Y, Kim M. How Strong is the Evidence for the Anxiolytic Efficacy of Lavender?: Systematic Review and Meta-analysis of Randomized Controlled Trials. Asian Nurs Res (Korean Soc Nurs Sci). 2019 Dec;13(5):295-305. doi: 10.1016/j.anr.2019.11.003. Epub 2019 Nov 16. PMID 31743795
- [Background] Maranets I, Kain ZN. Preoperative anxiety and intraoperative anesthetic requirements. Anesth Analg. 1999 Dec;89(6):1346-51. doi: 10.1097/00000539-199912000-00003. PMID 10589606